CLINICAL TRIAL: NCT01501643
Title: Non Invasive Positive Pressure Ventilation for Prevention of Acute Chest Syndrome in Sickle Cell Disease With Vaso-occlusive Crisis and Morphinic Treatment
Brief Title: Non Invasive Positive Pressure Ventilation for Prevention of Acute Chest Syndrome in Sickle Cell Disease
Acronym: VPACS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: decision of the promoter
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P091114
Record Dates: First submitted 2011-12-26; First posted 2011-12-29 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Sickle Cell-hemoglobin SS Disease; Vaso-occlusive Crisis
Keywords: Non invasive positive pressure ventilation; Spirometry; Acute chest syndrome; Sickle cell disease; Vaso-occlusive crisis
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Acute Chest Syndrome | interventions — Spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spirometry (Active Comparator): Spirometry
  Interventions: Device: Spirometry
- Non invasive positive pressure ventilation (Experimental): Non invasive positive pressure ventilation
  Interventions: Device: Non invasive positive pressure ventilation

INTERVENTIONS:
Device: Non invasive positive pressure ventilation — At least one hour every four hour but may be maintained more if the patient chooses to or is asleep with the machine on.
  Arms: Non invasive positive pressure ventilation
Device: Spirometry — Every two hours during the day with 10 maximum inspirations and at night if the patient is awake
  Arms: Spirometry

SUMMARY:
Acute chest syndrome is a severe respiratory complication of sickle cell disease.

The standard prevention of this dangerous complication is spirometry in wich patient is required to take deep breaths trough a little device several times a day. This treatment is compromised when pain in important or when the patient is asleep and cannot participate.

The investigators hypothesised that non invasive ventilation in wich patient have no effort to take might be a better prevention than spirometry and may improve pain and quality of sleep.

Children with vaso-occlusive crisis necessitating morphinic treatment will be randomly assigned with either spirometry or ventilation and the investigators will monitor for occurrence of acute chest syndrome, pain and quality of sleep.

DETAILED DESCRIPTION:
Acute chest syndrome is a severe complication of sickle cell disease. Several factors can contribute to this complication including infections, vaso-occlusive crisis, important pain that may give shortness of breath and morphinic treatments as they may cause hypoventilation.

The standard prevention of this dangerous complication is incentive spirometry in wich patient is required to take deep breaths trough a little device several times a day. This treatment is compromised when pain in important or when the patient is asleep and cannot participate.

In patients who have had surgery who have also pain and morphinic treatments, non invasive ventilation have proven a good option for preventing pulmonary complications.

Besides, our experience in non invasive ventilation for treatment of acute chest syndrome show a good tolerance and efficiency. It also seems to help with pain management.

The investigators hypothesised that non invasive ventilation in wich patient have no effort to take might be a better prevention than incentive spirometry and may improve pain and quality of sleep.

After informed consent, patients aged from 6 to 20 years old with SS or S-Beta sickle cell disease with vaso-occlusive crisis necessitating morphinic treatment hospitalised in intensive care unit in Necker Hospital for Sick Children (Paris) will be randomly assigned with either spirometry or ventilation. It is a monocentric study.

Patients with acute chest syndrome, oxygen needs, pneumonia or other condition requiring ventilation at presentation will not be included.

Spirometry will be realised through volumetric devices, every two hours during the day with 10 maximum inspirations and at night if the patient is awake.

Non invasive ventilation will be applied through a nasal mask with VS III machines from Resmed®, at least one hour every four hour but may be maintained more if the patient chooses to or is asleep with the machine on.

The investigators will monitor for occurrence of acute chest syndrome, pain, morphinic requirements, length of hospital stay, comfort, quality of sleep The treatment will be continued until morphinic treatment is stopped. The investigators intend to include 60 patients in each arm to show a difference of 25% in the occurrence of acute chest syndrome (primary judgement criteria).

Acute chest syndrome will be defined according to the criteria used by Vichinsky (Vichinsky, E. P. et al. Acute chest syndrome in sickle cell disease: clinical presentation and course. Cooperative Study of Sickle Cell Disease. Blood 89, 1787-1792 (1997) The investigators will aslo compare morphinic requirements, length of hospital stay and quality of sleep as secondary judgment criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patient with SS or S-Beta sickle cell disease aged more than 6 years old and less then 20 years old
* Hospitalised since less then 24 hours for severe vaso-occlusive crisis (either peripheric localisation or thoracic crisis) with morphinic requirements according to local pain management protocol
* With a signed informed consent from the patient or his legal representative if the patient is under 18 years old
* Benefiting of the French social security system

Exclusion Criteria:

* Patient that has already participated in the study
* Oxygen requirements, pneumonia, acute chest syndrome or other condition necessitating non invasive ventilation on admission
* No understanding of spirometry or ventilation techniques
* Other condition that forbid the use of non invasive ventilation or spirometry as defined by french consensus conference (2006) on non invasive ventilation

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Occurence of acute chest syndrome | up to 2 months at maximum (duration of hospitalization)

SECONDARY OUTCOMES:
Pain | up to 2 months at maximum (duration of hospitalization)
Morphinic requirements | up to 2 months at maximum (duration of hospitalization)
Length of hospital stay | up to 2 months at maximum (duration of hospitalization)
Comfort | up to 2 months at maximum (duration of hospitalization)
Quality of sleep | up to 2 months at maximum (duration of hospitalization)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Heilbronner, MD, PhD, Principal Investigator — Necker - Enfants Malades Hospital
Locations (1):
- Hôpital Necker - Enfants Malades Hospital, Paris, France